CLINICAL TRIAL: NCT05442749
Title: A Multicentric, Single Arm, Phase II Trial Assessing the Efficacy of Niraparib As First Line Therapy for Patients with Metastatic Homologous Repair-deficient Pancreatic Cancer
Brief Title: Niraparib As First Line Therapy with Metastatic Homologous Repair-deficient Pancreatic Cancer
Acronym: PARPi-PANC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study not feasible, patient accrual rate too low.
Sponsor: Centre Leon Berard (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET21-169
Record Dates: First submitted 2022-06-23; First posted 2022-07-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Niraparib (Experimental)
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Eligible patients will receive niraparib once daily, per os, continuously until loss of clinical benefit, unacceptable toxicity, death, patient or physician decision to withdraw, or pregnancy, whichever occurs first.
  300 mg/day, continuously for patients with TB >1.5- 3 ULN and/or ASAT/ALAT ≤5ULN.
  Or 200mg/day initial dosing for patients with TB >1.5 ULN and up to 3ULN and/or ASAT/ALAT > 2.5 ULN and up to 5 ULN with increase to 300mg/day if 1) liver safety lab tests improve to Grade 1 according to NCI criteria (based on total bilirubin and AST/ALT) with bilirubin < 1.5ULN) and 2) no grade >1 related AE are reported.

SUMMARY:
This trial is a single arm open-label, phase II aiming to assess the clinical activity of niraparib in chemotherapy-naïve biomarker-selected pancreatic cancer patients.

DETAILED DESCRIPTION:
This trial is a single arm open-label, phase II aiming to assess the clinical activity (objective response rate at week16 according to RECIST V1.1) of niraparib in chemotherapy-naïve biomarker-selected pancreatic cancer patients.

HR alterations must be confirmed before study drug start: only patients with mutation and/or rearrangement leading to inactivation in at least one of the following genes BARD1, BRCA1, BRCA2, BRIP1, FANCA, FANCD2, FANCL, MRE11, NBN, PALB2, PPP2R2A, RAD51B, RAD51C, RAD51D, RAD54L are eligible.

Eligible patients will receive niraparib once daily, per os, continuously until loss of clinical benefit, unacceptable toxicity, death, patient or physician decision to withdraw, or pregnancy, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient ≥18 years of age at time of informed consent form signature.
* Histologically proven advanced/metastatic PDAC not curable by surgery and/or definitive radiotherapy and not previously exposed to chemotherapy in advanced/metastatic setting. See Note in the full protocol
* Documented deleterious alteration resulting in inactivation in at least one of the following genes BARD1, BRCA1, BRCA2, BRIP1, FANCA, FANCD2, FANCL, MRE11, NBN, PALB2, PPP2R2A, RAD51B, RAD51C, RAD51D, RAD54L. See Notes in the full protocol
* Measurable disease at baseline according to RECIST V1.1 (See Section Appendix) See note in the full protocol
* Avaibility of a representative formalin-fixed paraffin-embedded (FFPE) sample of the primary or metastatic tumor tissue (resection or biopsy) with an associated pathology with the following quality/quantity control criteria: ≥30 % of tumor cells and a tumor surface area ≥ 5mm2.
* Optional - Tumor lesion visible by medical imaging and accessible to repeatable percutaneous or endoscopic sampling that permits core needle biopsy without unacceptable risk of a significant procedural complications, and suitable for retrieval of a minimum of 4 cores with a needle minimum diameter :16-gauge. See note in the full protocol.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 (See Section Appendix)
* Life expectancy > 16 weeks.
* Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 7 days prior to C1D1:

Parameters Laboratory Value

* Absolute neutrophil count ≥ 1.5 109/L
* Platelets ≥ 100 109/L
* Hemoglobin ≥ 9 g/dL (without transfusion within 7 d)
* Serum creatinine OR Creatinine clearance according to CKD-EPI ≥ 30 mL/min/1.73 m2 for patient with creatinine levels > 1.5 ULN

Serum total bilirubin :

300mg initial dosing: ≤ 1.5 x ULN (except for patients with Gilbert disease for whom a total serum bilirubin ≤ 3 x ULN is acceptable) OR Direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 x ULN 200mg initial dosing: up to 3 ULN

-- ASAT and ALAT : 300mg initial dosing: ≤ 2.5 x ULN (or up to 5 x ULN in case of liver metastasis or hepatic infiltration) 200mg initial dosing up to 5ULN

* Resting blood pressure systolic < 140 mmHg and diastolic <90 mmHg.
* Women patients of child-bearing potential are eligible, provided they have a negative serum or urine pregnancy test within 3 days prior to C1D1, and agrees to use a highly effective contraception (See section appendix) beginning signing the ICF to 6 months after the final dose of study drug.
* Fertile men must agree to use an effective method of contraception (See section appendix) during the study and for up to 3 months after the last dose of study drug and to not donate sperm during the same period.
* Patient should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures performed and should be able and willing to comply with study visits and procedures as per protocol.
* Patients must be covered by a medical insurance.

Exclusion Criteria:

* Patients not respecting the requirement for prior and concomitant treatment
* Inability to swallow capsules (bowel obstruction) or hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases. See notes in the full protocol
* Patients with other malignancy unless this malignancy is not expected to interfere with the evaluation of study endpoints (eg, basal or squamous cell carcinoma of the skin, in-situ carcinoma of the cervix, localized prostate cancer), or with no evidence of disease for ≥ 2 years.
* Any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
* History of severe allergic or other hypersensitivity reactions to any component of niraparib.
* Patients with:
* Active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) unless their HBV is stably controlled on nucleoside analogs (eg entecavir or tenofovir) which will be continued for the duration of the study. See note in the full protocol.
* Active hepatitis C. Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA, or
* HIV infection
* Prior organ or bone marrow transplant.
* Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Efficacy of niraparib in patients with HR-deficient pancreatic cancer | 16 weeks
  Objective response rate at Week 16 (ORR-16W) according to RECIST V1.1

SECONDARY OUTCOMES:
Disease control rate (DCR) | 16 weeks
  After 16 weeks of treatment (DRC-16W) according to RECIST V1.1
Best overall response Rate | At least 12 months following inclusion
  According to RECIST V1.1
Duration of response (DoR) | At least 12 months following inclusion
Progression Free survival (PFS) | At least 12 months following inclusion
Overall survival (OS) | At least 12 months following inclusion
Safety and tolerability of niraparib in pancreatic cancer patients | At least 12 months following inclusion
  incidence and severity of AEs (with severity determined according to NCI CTCAE v5.0)

OTHER OUTCOMES:
PD biomarkers of response and resistance to niraparib | At screening, cycle 3 day 1, cycle 5 day 1, cycle 7 day 1, (each cycle is 28 days) and at the end of study visit (within 30 days after last treatment administration)
  transcriptom profiling, HRD panel and HRD-signature (scarring / pattern), Dosing ctDNA & NGS/RNASeq

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Léon Bérard, Lyon, France